CLINICAL TRIAL: NCT03229122
Title: Japan CHARLOTTE: Characterizing the Cross-sectional Approach to Ovarian Cancer: Genetic Testing of BRCA
Brief Title: Characterizing the Cross-sectional Approach to Ovarian Cancer: Genetic Testing of BRCA
Acronym: CHARLOTTE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0816R00013
Record Dates: First submitted 2017-06-02; First posted 2017-07-25 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer, gBRCAm
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — From all the eligible subjects who have already attached the signature to the written informed consent, blood samples shall be collected. By using an assigned 10-mL EDTA-added blood collecting glass tube, 7 mL of the blood is sampled. The blood samples are to be recovered together with the specified test request form by Myriad and presence or absence of gBRCAm shall be centrally determined by US Myriad Genetics. Treatments of the samples, handling procedures and recovery methods are precisely described on the testing manual.
  The physician responsible for institutional study has the responsibility to notify the gBRCAm results to all the patients who underwent the tests. However, this responsibility needs not to be observed if the patients themselves refuse such a notification about gBRCAm test results. This responsibility shall be assumed by the physician responsible for institutional study in each participating institute.
  Incidentally, the genetic test results of the patients should
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The multi-centered, cross-sectional investigations shall be conducted in this study with the objective of identifying the ownership ratio of gBRCAm on the newly diagnosed patients with epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer in Japan.

DETAILED DESCRIPTION:
This multi-centered, cooperative and epidemiological observation study is so designed to investigate the ownership ratio of gBRCAm in the newly diagnosed patients with epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer because such a ratio has not yet been adequately clarified in Japan.

The newly diagnosed eligible patients with epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer shall be asked to participate in this study in order of diagnosis. After obtaining their consents by the written informed consent following appropriate explanation, investigations about the demographic information including the cancer family history shall be performed. Subsequently, blood is collected for investigation about gBRCAm. In addition, histological classification shall be conducted based on the resected tumor tissues.

ELIGIBILITY:
Inclusion Criteria:

For registration to this study, all of the following criteria should be satisfied:

1. The subject can attach the signature to the Informed Consent Form (ICF), besides having his/her intention to put the signature.
2. Female Japanese at more than 20 years of age
3. The newly diagnosed patients whose epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer is histologically confirmed as FIGO from the subject to obtain their utmost understandings. Limited to histopathological diagnosis based on resected tumor specimens (except the cytodiagnosis by ascites paracentesis).
4. The histopathological specimens can be submitted to the central pathological judgment.
5. Within 60 days after diagnosis of epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer, the patient's written consent has been obtained.

Exclusion Criteria:

* The subjects who coincide any of the following exclusion criteria are designated to be ineligible:

  1. In case of the subjects who are diagnosed to have acute or chronic physical or severe mental diseases except cancer, and about whom the attending responsible physician makes judgement to say that participation of these subjects would possibly increase the risks or would probably disturb the interpretation of the study results.
  2. In case of the subjects whose registration for the study is judged by the attending responsible physician as inappropriate.

Ages: 20 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female Japanese at more than 20 years of age
Study Population: The newly diagnosed patients with epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 446 (Estimated)
Dates: Start 2016-12-26 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the ownership ratio of gBRCAm in the newly diagnosed patients with epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer in Japan. | Baseline
  To be evaluated based on laboratory test.

SECONDARY OUTCOMES:
Ownership ratio of gBRCAm when stratified according to the patients' demographics | Baseline
  To be evaluated by laboratory test
Evaluation of the satisfaction levels of the patients toward explanation about the BRCA genetic testing | Baseline
  To be evaluated by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Toru Sugiyama, MD, Principal Investigator — Iwate Medical University; Daisuke Aoki, MD, Study Director — Keio University; Takayuki Enomoto, MD. PhD., Study Director — School of Medicine, Niigata University; Nobuhiro Takeshima, MD., Study Director — The Cancer Institute Hospital Of JFCR.; Junzo Kigawa, MD, PhD, Study Director — The Matsue City Hospital; Yo Watanabe, Study Director — The Tohoku Medical and Pharmaceutical University; Masami Arai, MD. PhD., Study Director — The Cancer Institute Hospital Of JFCR.
Locations (35):
- Japan (35):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Izumo
  - Research Site, Kanagawa
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Maebashi
  - Research Site, Matsuyama
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Morioka
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Tōon
  - Research Site, Yamagata

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4549&filename=Study_report_synopsis_D0816R00013_redacted.pdf